CLINICAL TRIAL: NCT04569461
Title: Trimodality Approach of Low Dose iOnizing Radiation With or Without Neoadjuvant Pembrolizumab and Prostatectomy for Men With Intermediate/High Risk Prostate Cancer (TALON)
Acronym: TALON
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinuation of funding
Sponsor: Duke University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103396
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; KEYTRUDA; pembrolizumab; prostatectomy; localized prostate cancer; prostate radiation; low dose prostate radiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: pembrolizumab, low dose prostate radiation and prostatectomy (Experimental): Participants in Arm A will receive:
  * Pembrolizumab 400 mg intravenously every 6 weeks for 9 cycles.
  * Low dose prostate radiation of one dose of 2 Gy to the prostate and seminal vesicles
  * Prostatectomy as part of the routine care for their cancer
  Interventions: Drug: pembrolizumab; Radiation: Low dose prostate radiation; Procedure: Radical Prostatectomy
- Arm B: Low dose prostate radiation and prostatectomy (Experimental): Participants in Arm B will receive:
  * Low dose prostate radiation of one dose of 2 Gy to the prostate and seminal vesicles
  * Prostatectomy as part of the routine care for their cancer
  Interventions: Radiation: Low dose prostate radiation; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: pembrolizumab — 400 mg of pembrolizumab (KEYTRUDA) will be given by IV every 6 weeks for 9 cycles, for approximately one year of study drug administration.
  Other Names: KEYTRUDA
  Arms: Arm A: pembrolizumab, low dose prostate radiation and prostatectomy
Radiation: Low dose prostate radiation — A single dose of 2 Gy of radiation will be given to the prostate and seminal vesicles on approximately Week 7 for Arm A and approximately 2 weeks prior to the prostatectomy for Arm B.
Procedure: Radical Prostatectomy — Robotic assisted laparoscopic prostatectomy (RALP) surgery will be performed at approximately Week 9 for Arm A and approximately 2 weeks after the low dose prostate radiation for Arm B. This surgery is part of the participants routine medical care.
  Other Names: Robotic assisted laparoscopic prostatectomy (RALP)

SUMMARY:
This study will enroll prostate cancer patients with an unfavorable intermediate- or high-risk diagnosis. The purpose of this study is to determine whether a regimen of pembrolizumab and low dose prostate radiation or low dose prostate radiation alone prior to a prostatectomy affects cells of the immune system and if it is a safe option for this stage of prostate cancer. Participants will be randomized 1:1 (like flipping a coin) to receive pembrolizumab, low dose prostate radiation and a prostatectomy or low dose prostate radiation and a prostatectomy. Pembrolizumab is an investigational drug that increases the ability of the immune system to kill tumor cells. Low dose radiation can alter the way tumor cells look to the immune cells. For example, the immune cells may express different proteins that make them more susceptible to immune cell killing or the structure of the tumor may be altered to allow the immune cells to infiltrate the tumor more thoroughly. The prostate tissue collected from the prostatectomy will be analyzed for differences in pathology and local immune cell infiltration, and participants will be followed for 2 years to watch for prostate specific antigen (PSA) recurrence and prostate cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document.
2. Age ≥ 18 years
3. Histologic evidence of adenocarcinoma of the prostate who are deemed candidates for radical prostatectomy. Variants such as neuroendocrine components or ductal carcinoma are allowed. Pure small cell carcinoma is not allowed.
4. At least one unfavorable intermediate or high risk factors or classified as high risk clinically localized disease as defined by NCCN guidelines:

   a. High risk: At least one of the following: i. cT3a disease ii. Gleason sum of 8, 9 or 10 iii. PSA ≥ 20 ng/ml

   b. At least one of the following unfavorable intermediate risk factors:: i. cT2b or cT2c disease ii. Grade group 3 iii. PSA 10-20 ng/ml iv. Grade group 2 and 50% or greater prostate biopsies positive for cancer
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (See Appendix A)
6. Adequate normal organ and marrow function as defined below by the following criteria within 10 days prior to first dose of study treatment.:

   1. Hemoglobin ≥ 9.0 g/dL
   2. Absolute neutrophil count (ANC ≥1.5 x 10^9/L)
   3. Platelet count ≥100 x 10^9/L
   4. Serum bilirubin ≤ 1.5 x Institutional Upper Limit of Normal (ULN)
   5. AST/SGOT and ALT/SGPT ≤ 2.5 x ULN
   6. Measured creatinine clearance (CL) >50 mL/min

8. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. History of or known bone, brain, visceral, or soft tissue metastasis, including lymph nodes based on standard of care imaging with CT or pelvic MRI showing no LNs greater than 1.5cm and bone scan showing no evidence of bone metastasis.
2. Prior pelvic radiation or prostate cryotherapy or high-intensity focused ultrasound (HIFU)
3. Any prior treatment with PD-1 or PD-L1 checkpoint inhibitors or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137, PD-L2).
4. Has received an investigational agent (or used an investigational device) within 4 weeks prior to study intervention administration.

   a. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
5. Prior therapy for prostate cancer

   a. Exceptions: Previous alpha-reductase inhibitor use allowed IF patient has not been taking for at least 30 days prior to study treatment initiation, OR if alpha reductase inhibitor was not used as a primary treatment of prostate cancer and the PSA on alpha-reductase inhibitor remains within eligibility when doubled.
6. Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
7. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid).
8. Presence of a condition requiring chronic steroid use (equivalent to >10 mg of prednisone daily) or other immunosuppressive drugs (i.e., for organ transplant). The following are exceptions to this criterion:

   1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   2. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
9. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
10. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of investigational product (IP) and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease
11. History of allogenic stem cell transplant
12. History of active primary immunodeficiency
13. Known history of human immunodeficiency virus
14. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
15. Has not adequately recovered from major surgery or has ongoing surgical complications.
16. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
17. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
18. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
19. Any condition which, in the opinion of the investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Total number of CD8+ T-cells in prostatectomy samples | Prostatectomy (Week 7 for Arm A, Week 3 for Arm B)
  Total number of CD8+ T-cell profiles in prostate tumor samples removed by RALP in men treated with preoperative low dose prostate radiation (LDPR) alone or with preoperative pembrolizumab.
Location of CD8+ T-cells in prostatectomy samples | Prostatectomy (Week 7 for Arm A, Week 3 for Arm B)
  Description of location of CD8+ T-cell profiles of prostate tumor samples removed by RALP in men treated with preoperative low dose prostate radiation (LDPR) alone or with preoperative pembrolizumab.
Characteristics of CD8+ T-cells in prostatectomy samples | Prostatectomy (Week 7 for Arm A, Week 3 for Arm B)
  Description of Characteristics of CD8+ T-cell profiles of prostate tumor samples removed by RALP in men treated with preoperative low dose prostate radiation (LDPR) alone or with preoperative pembrolizumab.

SECONDARY OUTCOMES:
Acute safety profile | 30 days after prostatectomy
  Description of the acute (30 day) safety profile of participants receiving low dose prostate radiation pre-operatively with or without pembrolizumab
Long term safety profile | 2 years after prostatectomy
  Description of the long term (2 year) safety profile of participants receiving low dose prostate radiation pre-operatively with or without pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Daniel George, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No